CLINICAL TRIAL: NCT03596931
Title: Prior Statin Use and Risk of Heart Failure, Acute Lung Edema and Malignant Arrhythmia in Indonesian Post-Acute Coronary Syndrome Patients
Brief Title: Prior Statin Use and Risk of CHF, ALO and Malignant Arrhythmia in Indonesian Post-Acute Coronary Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Tarumanagara University (Other)
Collaborators: Cengkareng General Hospital (Other)
Responsible Party: Principal Investigator, Angela Felicia Sunjaya, Co Principal Investigator, Tarumanagara University
Other Study IDs: APS004
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndrome; Acute Pulmonary Edema; Arrhythmias, Cardiac; Heart Failure
Keywords: acute coronary syndrome; statin; acute pulmonary edema; malignant arrhythmia; heart failure
MeSH Terms: conditions — Acute Coronary Syndrome; Arrhythmias, Cardiac; Heart Failure | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Cardiovascular Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin: History of statin use prior to Acute Coronary Syndrome
  Interventions: Drug: Statins (Cardiovascular Agents)
- Non-Statin: No documented history of statin use prior to Acute Coronary Syndrome

INTERVENTIONS:
Drug: Statins (Cardiovascular Agents) — Prescribed with statins
  Groups: Statin

SUMMARY:
This study aims to evaluate the effect of statin for primary prevention, towards lowering the incidence of heart failure, acute lung edema, malignant arrhythmia and death in ACS patients.

DETAILED DESCRIPTION:
Adult patients (≥ 18 years of age) with acute coronary syndrome which are diagnosed under ICD-10 coding of I24.9 without a prior history of heart failure, acute lung edema and arrhythmia were included in this study. The inclusion criteria are patients with primary diagnosis of I24.9 and with a complete record of prior medical and treatment history, electrocardiographic findings, cardiac marker results and outcomes. Participants were grouped into 2 groups - statin and non-statin based on prior history of statin use prior to ACS. Diagnosis of ACS was made based on clinical, electrocardiographic and cardiac marker findings found in the medical record.

Data such as age, sex, ethnic, education, prior medical and treatment history, electrocardiographic and cardiac enzyme results as well as outcomes were collected from the patients' medical records. Outcomes of interest were defined as either concomitant heart failure, acute lung edema, malignant arrhythmia, mortality or combinations of them as diagnosed in the medical records. Heart failure is defined based on echocardiographic findings from the medical records. Acute Lung Edema is defined based on medical records or reported clinical findings of lung edema - rhonchi reported in 1/3 of the lungs with oxygen saturation <90%. Whereas malignant arrhythmia is defined as the presence of ventricular tachycardia (VT) or ventricular fibrillation (VF).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Coronary Syndrome
* Presence of detail on statin prescription history

Exclusion Criteria:

* History of heart failure, acute lung edema and arrhythmia
* Unavailability of electrocardiographic findings, cardiac marker results
* Incomplete records of prior medical and treatment history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) with acute coronary syndrome which are diagnosed under ICD-10 coding of I24.9 without a prior history of heart failure, acute lung edema and arrhythmia.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Heart Failure | Through study completion, an average of 1 year
  Based on echocardiographic findings from the medical records
Malignant Arrhythmia | Through study completion, an average of 1 year
  Presence of ventricular tachycardia (VT) or ventricular fibrillation (VF)
Acute Lung Edema | Through study completion, an average of 1 year
  Based on medical records or reported clinical findings of lung edema - rhonchi reported in 1/3 of the lungs with oxygen saturation <90%.

CONTACTS AND LOCATIONS:
Overall Officials: Andria Priyana, MD, FIHA, Study Chair — Department of Cardiology, Faculty of Medicine, Tarumanagara University; Angela F Sunjaya, Principal Investigator — Tarumanagara University; Anthony P Sunjaya, Principal Investigator — Tarumanagara University
Locations (1):
- Cengkareng General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided